CLINICAL TRIAL: NCT05562609
Title: Tranexamic Acid by the Intramuscular or Intravenous Route for the Prevention of Postpartum Haemorrhage in Women At Increased Risk: a Randomised, Double-blind, Placebo-controlled Trial
Brief Title: Tranexamic Acid to Prevent Heavy Bleeding After Childbirth in Women At Higher Risk
Acronym: I'M-WOMAN
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: UNITAID (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IMWOMAN
Record Dates: First submitted 2022-09-27; First posted 2022-10-03 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Postpartum Hemorrhage
Keywords: tranexamic acid; postpartum haemorrhage; bleeding; pregnancy; antifibrinolytic; intramuscular
MeSH Terms: conditions — Postpartum Hemorrhage; Hemorrhage | interventions — Tranexamic Acid; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Masking done by an independent clinical trials supply company. It will involve the removal of the original manufacturer's label and replacement with the clinical trial label bearing the randomisation number, which will be used as the pack identification. Apart from the randomisation number, all pack label texts and ampoules will be identical for each arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intramuscular TXA (Experimental): 1g TXA as 2 x 5 ml IM injections (100mg/ml) and slow IV injection of placebo (1 x 10 ml of 0.9% sodium chloride)
  Interventions: Drug: Tranexamic acid; Other: Placebo
- Intravenous TXA (Active Comparator): 1g TXA by slow IV injection and 2 x 5 ml IM injections of placebo
  Interventions: Drug: Tranexamic acid; Other: Placebo
- Placebo (Placebo Comparator): Placebo by 1 x slow 10ml IV injection and 2 x 5 ml IM injections
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Tranexamic acid — Ampoules and packaging for all arms will be identical in appearance.
  Other Names: Cyklokapron
  Arms: Intramuscular TXA; Intravenous TXA
Other: Placebo — Ampoules and packaging for all arms will be identical in appearance.
  Other Names: (Sodium Chloride 0.9%)

SUMMARY:
Heavy bleeding after childbirth, known as a postpartum haemorrhage (PPH), causes about 70,000 maternal deaths every year. Tranexamic acid (TXA) is a lifesaving treatment for women with PPH. The I'M WOMAN trial is a research study to see whether giving TXA just before childbirth will stop women developing PPH. The trial will assess the effects of intramuscular (IM) and intravenous (IV) tranexamic acid on PPH, side effects and other important maternal health outcomes.

DETAILED DESCRIPTION:
Postpartum haemorrhage (PPH) causes about 70,000 maternal deaths every year. Tranexamic acid (TXA) is a lifesaving treatment for women with PPH. The WOMAN trial recruited over 20,000 women with PPH and found that intravenous (IV) TXA given soon after PPH onset, reduces bleeding deaths by about a third. Early TXA also reduces blood loss in surgery and death due to bleeding after traumatic injury. The World Health Organization recommends that all women with PPH should receive TXA as a first line treatment.

TXA is more effective when given soon after the bleeding starts. Every fifteen minute delay reduces the survival benefit by about 10%. This suggests that giving TXA around the time of childbirth might prevent PPH. Although several clinical trials have examined the effectiveness of TXA for the prevention of PPH, the results are inconclusive. Trials of tranexamic acid for PPH prevention give the trial treatment after cord clamping, which may be too late to prevent bad bleeding in some women, as bleeding tends to happen soon after childbirth. Because PPH only affects a small proportion of births, the healthcare community need good evidence on the balance of benefits and harms in this population before using TXA to prevent PPH.

The I'M WOMAN trial will evaluate the effects of TXA for PPH prevention in women with one or more risk factors for PPH having a vaginal or caesarean birth. The trial will also evaluate the effect of the route of TXA administration. TXA is usually given by slow IV injection. However, recent research shows that TXA is well tolerated and rapidly absorbed after IM injection, achieving therapeutic blood levels within minutes of injection. There may be fewer side effects with IM TXA because peak blood concentrations are lower than with the IV route, as well as practical advantages.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 years or older who are admitted to hospital to give birth vaginally or by caesarean section, who have one or more known risk factors for PPH

Exclusion Criteria:

* Women who have a clear indication or contraindication for TXA

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30000 (Estimated)
Dates: Start 2024-04-22 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Risk of Postpartum haemorrhage | within 24 hours of childbirth
  Clinical assessment: This may be an estimated blood loss of more than 500 mL in vaginal births or more than 1000 ml in caesarean births, or any blood loss sufficient to compromise haemodynamic stability. Haemodynamic instability is based on clinical judgement and assessed using clinical signs (low systolic blood pressure, tachycardia, reduced urine output)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Brenner, Study Director — London School oh Hygiene and Tropical Medicine
Locations (1):
- Mbeya Regional Referral Hospital, Mbeya, Tanzania

IPD SHARING:
Plan to Share IPD: Yes
The investigators are committed to sharing data for ethical research with justified scientific objectives. Until all planned analyses are completed by the LSHTM CTU Global Health Trials Group, data will be shared through a controlled access approach whereby researchers can make formal applications for data sharing. Afterwards, the anonymised dataset will be shared via the LSHTM CTU Global Health Trials Group data sharing platform at freebird.lshtm.ac.uk. All trial materials including training materials, CRFs and Protocol will be made available on the trial website and team YouTube channel.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Once all planned analyses are completed by the LSHTM CTU Global Health Trials Group following trial completion. Data will be shared indefinitely.
Access Criteria: As above
URL: http://freebird.lshtm.ac.uk

REFERENCES:
- [Derived] Larson NJ, Mergoum AM, Dries DJ, Cook A, Blondeau B, Rogers FB. THE ROLE OF TRANEXAMIC ACID IN POSTPARTUM HEMORRHAGE: A NARRATIVE REVIEW. Shock. 2024 Nov 1;62(5):620-627. doi: 10.1097/SHK.0000000000002455. Epub 2024 Aug 20. PMID 39162220
- [Derived] Brenner A, Shakur-Still H, Chaudhri R, Muganyizi P, Olayemi O, Arribas M, Kayani A, Javid K, Bello A, Roberts I; I'M WOMAN Trial Collaborative Group. Tranexamic acid by the intramuscular or intravenous route for the prevention of postpartum haemorrhage in women at increased risk: a randomised placebo-controlled trial (I'M WOMAN). Trials. 2023 Dec 3;24(1):782. doi: 10.1186/s13063-023-07687-1. PMID 38044460